CLINICAL TRIAL: NCT07229560
Title: The Effect of Itraconazole on the Pharmacokinetics of Orally Administered HRS-8080 in Healthy Participants: A Single-Center, Single-Arm, Open-Label, Fixed-Sequence Study
Brief Title: A Trial of Itraconazole Effect on HRS-8080 Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-105
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-8080 Tablets and Itraconazole Capsules Group (Experimental)
  Interventions: Drug: HRS-8080 Tablet; Drug: Itraconazole Capsule

INTERVENTIONS:
Drug: HRS-8080 Tablet — HRS-8080 tablet, specified dose on specified days.
Drug: Itraconazole Capsule — Itraconazole capsule, specified dose on specified days.

SUMMARY:
This is a phase I study to evaluate the effect of Itraconazole on the pharmacokinetics of HRS-8080 in healthy participants and the safety of HRS-8080 administered alone and in combination with Itraconazole in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-55 years;
2. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 19-28 kg/m2;
3. Normal or no clinically significant medical history, ECGs, vital signs and laboratory tests;
4. Take contraception.

Exclusion Criteria:

1. Any serious clinical diseases or medical history or diseases that affect the absorption, metabolism and/or excretion of the study drug;
2. Severe infection, severe trauma or major surgery;
3. Any medications in the two weeks before screening or baseline period;
4. History of blood donation or severe blood loss;
5. Have been vaccinated within 3 months before the screening or baseline period;
6. History of smoking or excessive alcohol or drug abuse;
7. History of excessive amounts of tea, coffee or caffeinated beverages, special foods; or have special dietary requirements;
8. Other situations in which the researcher judges unsuitable.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-11-26 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of HRS-8080. | From Day 1 to Day 11.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) of HRS-8080. | From Day 1 to Day 11.
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) of HRS-8080. | From Day 1 to Day 11.

SECONDARY OUTCOMES:
Time to maximum plasma concentration (Tmax) of HRS-8080. | From Day 1 to Day 11.
Terminal elimination half-life (t1/2) of HRS-8080. | From Day 1 to Day 11.
Apparent volume of distribution (Vz/F) of HRS-8080. | From Day 1 to Day 11.
Clearance (CL/F) of HRS-8080. | From Day 1 to Day 11.
Adverse events (AEs). | From Day 1 to Day 17.
Serious adverse events (SAEs). | From Day 1 to Day 17.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided